CLINICAL TRIAL: NCT03521804
Title: A Single-Arm Study to Assess the Safety and Efficacy of the SoundBite™ Crossing System With ACTIVE Wire in Coronary Chronic Total Occlusions (the ACTIVE Trial).
Brief Title: Safety and Efficacy Study of the SoundBite™ Crossing System With ACTIVE Wire in Coronary CTOs.
Acronym: ACTIVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: SoundBite Medical Solutions, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAP-COR-2018-01
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion; coronary; SoundBite™ Crossing System; CTO; distal cap; true lumen; Active wire; Device; Procedure; Stenosis; CAD; Coronary Artery Disease
MeSH Terms: conditions — Constriction, Pathologic; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SoundBite™ Crossing System-Coronary (Other): Crossing of coronary chronic total occlusions.
  Interventions: Device: SoundBite™ Crossing System Active Wire 14

INTERVENTIONS:
Device: SoundBite™ Crossing System Active Wire 14 — Successful crossing of the CTO into the true arterial lumen distal to the occlusion, following use of the SoundBite™ Crossing Wire during the procedure and using antegrade only approach. An antegrade only approach may involve Antegrade Dissection Re-Entry (ADR) with or without the use of specialized devices (i.e. Stingray). The absence of successful retrograde crossing of a collateral will still be considered an antegrade only approach.

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the SoundBite™ Crossing System - Coronary (SCS-C) in a subject population with chronic coronary artery disease including Chronic Total Occlusion (CTO).

DETAILED DESCRIPTION:
The study is intended to demonstrate that the SoundBite™ Crossing System - Coronary can facilitate the passage of either 1) devices intended to treat a CTO or 2) guidewires or additional crossing devices into the true lumen distal to the CTO.

SoundBite™ Crossing System - Coronary, which consists of a re-usable console and a disposable device (ACTIVE Wire).

The SoundBite™ Crossing System - Coronary is intended to facilitate passage of a guidewire or therapeutic devices through a coronary artery Chronic Total Occlusion.

This is a prospective, multi-center, multinational, single-arm, phased clinical study intended to provide pivotal data for device approval.

ELIGIBILITY:
General inclusion Criteria

1. Subject planned to undergo clinically driven percutaneous coronary intervention (PCI) targeting a single CTO. Clinical justification of a CTO PCI includes anginal symptoms, dyspnea or left ventricular dysfunction presumed or documented to be the result of ischemia in the CTO territory.
2. PCI procedure is planned to be performed with a wire based antegrade primary strategy.
3. Subject is ≥ 18 years old.
4. Subject is able and willing to provide written informed consent prior to study procedure.

Angiographic Inclusion Criteria All angiographic inclusion criteria shall be documented at time of index procedure. Angiographic inclusion criteria are assessed at the site and determined by the site investigator.

1. Target CTO is in a native coronary artery and demonstrates TIMI flow grade 0.
2. Target CTO is presumed documented angiographically to be greater than 3 months old.
3. Target CTO length is visually estimated to be ≥ 5mm.
4. Target reference vessel diameter ≥ 2.5mm.
5. Target CTO shows calcification.
6. Target CTO has a positive tap test, which correspond to the inability to penetrate the cap by visual estimate using a polymer-jacketed or enhanced tip stiffness (>1.5 gm) coronary guidewire manipulated with the intention to cross the occlusion for at least 60 seconds of fluoroscopy time after initial guidewire-cap contact. The tap test is intended to confirm the chronicity of the lesion and rule out acute or sub-acute occlusions that will likely be crossed with such simple wire maneuvers.

General Exclusion Criteria

1. Life expectancy < 1 year.
2. Hypersensitivity or contraindication to aspirin, P2Y12 platelet receptor inhibitors, heparin or radiographic contrast agents which cannot be adequately pre-medicated, desensitized or where no alternative is available.
3. Target occlusion has an iatrogenic dissection that occurred within the past 3 months.
4. Subject has received ≥5 Gy exposure to the chest within 3 months.
5. Subject has known elevated cardiac biomarkers (CK-MB or cTn) within 30 days prior to index procedure.
6. Left ventricular ejection fraction less than 20%.
7. Severe aortic or mitral valve disease.
8. Planned left ventricular (LV) support device during CTO PCI.
9. History of bleeding diatheses, coagulopathy.
10. Recent (within 6 months prior to index procedure) stroke or transient ischemic attack (TIA).
11. Recent (within 6 months prior to index procedure) significant gastrointestinal (GI) bleeding.
12. Planned additional coronary or valvular percutaneous or surgical intervention scheduled within 30 days after index procedure.
13. Requires emergent or urgent PCI.
14. Positive pregnancy test result in women of child bearing potential or is breast-feeding.
15. Current participation in another investigational drug or device trial.
16. Other medical illnesses that may cause the subject to be non- compliant with the protocol or confound data interpretation.
17. Estimated Glomerular Filtration Rate (GFR) below 25 ml/min and not yet on dialysis.
18. Evidence of clinical instability (e.g., hemodynamic instability, sustained tachyarrhythmias, cardiogenic shock).

Angiographic Exclusion Criteria All angiographic inclusion criteria shall be documented at time of index procedure. Angiographic exclusion criteria are assessed at the site and determined by the site investigator.

1. Target CTO is in an unprotected left main.
2. No angiographically visible collateral flow to the target vessel distal to the occlusion, from ipsilateral or contralateral collaterals.
3. Vessel tortuosity proximal to, or within, body of target occlusion which, in the opinion of the investigator, is not amenable to advancement of a microcatheter or SoundBite™ Crossing System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Device success | Day 1
  Device Success defined as: Successful antegrade crossing of the CTO into the true arterial lumen distal to the occlusion following advancement of at least 3 mm of the Soundbite(TM) Crossing System into any segment as assessed by the core angiographic laboratory. An antegrade only approach may involve Antegrade Dissection Re-Entry (ADR) with or without the use of specialized devices (e.g. Stingray); absence of successful retrograde crossing of a collateral will still be considered an antegrade only approach.
Freedom from the composite SoundBite™ Crossing System related MAEs | 48 hours or until discharge
  Freedom from the composite SoundBite™ Crossing System related major adverse events (MAEs) at 48 hours or hospital discharge (whichever occurs first) post procedure, as per Clinical Events Committee (CEC) adjudication, defined as:
  * Cardiovascular related deaths
  * Myocardial Infarction (Primary definition of clinically relevant post procedure MI from SCAI (1).
  * Coronary Artery Perforation requiring treatment
  * Unscheduled cardiac surgery anytime between enrollment to completion of the study.
  * Intra-procedure stroke
  * Radiation exposure ≥ 8 Gy

SECONDARY OUTCOMES:
Overall Device Success | Day 1
  Successful crossing of the CTO, following use of the SoundBite™ Crossing Wire during the procedure including antegrade or retrograde approach.
Technical Success | Day 1
  Successful antegrade or retrograde crossing of the CTO into the true arterial lumen following advancement of at least 3 mm of the Soundbite Crossing System into the proximal segment as assessed by the core angiographic laboratory, with stent implantation and restoration of TIMI 3 flow, with less than 30% residual stenosis
Procedural Success | Day 1
  Achievement of Technical Success with freedom from In-Hospital device related MAEs per CEC adjudication.
Clinical Success: | 30 days post-procedure
  Achievement of Procedural Success with freedom from device related MAEs through 48 hours or hospital discharge and 30 days post index procedure.
Freedom from SoundBite™ Crossing System related MAE | 30 days post-procedure
  Freedom from SoundBite™ Crossing System related MAE assessed through 30 days post-index procedure, per CEC adjudication. Secondary MAE analysis employing the Third Universal consensus definition of Myocardial Infarction (MI)

CONTACTS AND LOCATIONS:
Locations (5):
- Columbia University Medical Center/NYPH, New York, New York, United States
- Canada (4):
  - ICM - Institut de Cardiologie de Montreal, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - MUHC- McGill University Health Centre, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec - IUCPQ, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No